CLINICAL TRIAL: NCT01072669
Title: Evaluation of the Effect of Ambrisentan on Digital Microvascular Flow in Patients With Systemic Sclerosis Using Laser Doppler Perfusion Imaging
Brief Title: Efficacy of Ambrisentan in Limited Scleroderma Patients in Improving Blood Flow to Hands or Feet
Acronym: ambrisentan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soumya Chatterjee (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Soumya Chatterjee, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: nbose2010
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Ischemia
Keywords: Ambrisentan increases digital micro-vascular flow (measured by LDPI) in patients with Raynaud's phenomenon (RP) and digital ischemia secondary to SSc.
MeSH Terms: conditions — Ischemia | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ambrisentan (Active Comparator): drug arm
  use of ambrisentan in limited scleroderma patients with raynaud's to evaluate digital microvascular flow
  Interventions: Drug: ambrisentan
- sugar pill (Placebo Comparator): those getting sugar pill to evaluate if the active drug improves digital microvascular flow in limited scleroderma patients
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — Subjects will receive ambrisentan 5 mg orally once daily or identical placebo pills for the first 4 weeks and then increased to ambrisentan 10mg once daily[if the lower dose is tolerated] or identical placebo pills for the rest of the study. They will be instructed to take the 5mg/pink pills for 4 weeks and then switch to 10mg /red pills unless they are having any drug related side effects or concerns. There will be no routine visit planned at 4 weeks to assess drug tolerance unless a complication arises. Adherence to treatment will be assessed by pill counting at each follow up visit. Follow up digital blood flow measurements will be obtained with LDPI at 1 week and at 3 months, where the same protocol (as that in the initial visit) will be followed.
  Other Names: Letairis

SUMMARY:
The purpose of this study is to investigate the effectiveness of a drug called ambrisentan, approved by the FDA for use in pulmonary hypertension (a condition where there is increased pressure in the right side of the heart) in scleroderma patients, to see if this medicine may be beneficial in relieving and/or preventing Raynaud's flares in you and other patients like you. This medicine may have some short-term and long-term benefits in persons with scleroderma

DETAILED DESCRIPTION:
Baseline screening-we will screen you with a baseline review of your history, medications and lab values and you will need to get blood drawn for hemoglobin level, liver function panel and blood pregnancy test for females in child bearing age group. Women are advised strongly to use 2 reliable forms of contraception while in this study unless you have had tubal ligation or intrauterine device placement.

You are advised to stop taking medications like nitrates (like nitroglycerin), calcium channel blockers (like nifedipine or amlodipine), angiotensin converting enzyme inhibitors (like lisinopril or enalapril or captopril), angiotensin receptor blockers (like valsartan or candesartan) or phosphodiesterase inhibitors (like Viagra or Revatio) at least 1 week prior to you coming for the first visit for the study and abstain from them during study period unless absolutely necessary.

Please avoid caffeine, smoking and over the counter cold remedies at least 2 days prior to the first visit and during the study period.

You will be asked to go to the Clinical Research Unit( CRU) located on M 51 in Cleveland Clinic main campus to partake in the study and will go back there for subsequent visits at 1 week and then at 12 weeks after having started the study.

This is a placebo-controlled randomized trial where 15 patients will get the active medication and the other 5 will get a placebo (pill with no active ingredient but not harmful to you in any way). This means you have a 3 in 4 (75%) chance of getting the active medication (ambrisentan) versus the placebo- both pills will look exactly the same. This process is called "randomization" and is similar to flipping a coin. The patients getting the active medication versus placebo will be randomly selected by the computer; the medications will be distributed by the central pharmacy and sent to the nurses on CRU and given to you on your first visit to the CRU. No one will know who received the active medication versus the placebo till the study ends and the data is analyzed.

Those getting the active medicine ambrisentan will initially get a dose of 5mg by mouth daily and then the dose will be increased to 10mg by mouth daily after 4 weeks if the medicine is well tolerated. This will be done by the computer for randomization/selection and the pharmacist for drug dispensing. If you experience any side effects, please contact us for further advice. You will be evaluated each visit by the nurses at weeks 0, 1 and 12 for any drug related problems. We will be monitoring the routine scheduled blood work results to make sure you do not develop any drug related problems which can be detected on blood work.

A machine called the 'Laser Doppler Perfusion Imaging' machine will be used at each of your visits to the CRU at weeks 0, 1 and 12. This machine uses simple laser beams and will scan the top part of your non-dominant hand (the left hand for most people) to measure the blood flow through the blood vessels there when your hand is at room temperature (around 77'F) and when it has been cooled to 50'F for 2 minutes with the help of a cold flask. This is a safe and simple technique and does not involve any radiation exposure.

You will also be asked to fill out 3 questionnaires at each of visits (week 0, 1 and 12) to the CRU-these have some simple questions regarding your degree of pain, severity of Raynaud's symptoms and the effect of scleroderma in your day-to-day functioning.

Please budget at least 1-2 hours for your initial visit (week 0) to the CRU and then 1 hour for your visits at 1 week and 12 weeks to the CRU.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have limited scleroderma with disease duration <7 years and should satisfy American College of Rheumatology criteria for diagnosis.9;
* 10 Raynaud's phenomenon would be defined as episodic, bilateral, digital color changes (at least 2 out of 3 possible phases:

  * pallor, cyanosis, rubor),
  * provoked by cold or emotional stress.
* Subjects should be between 18 and 70 years of age and be able to give informed consent.

Exclusion Criteria:

* (a) current tobacco users,
* (b) advanced cardiopulmonary disease,
* (c) clinically unstable patient,
* (d) presence of active digital ulcers or prior history of digital ulcers which led to scarring or significant pitting of digits in the area of interest(presence of ulcers or pits would interfere with measurement of blood flow by LDPI),
* (e) pregnancy (class X in pregnancy) or unable to use two reliable forms of contraception during the study if patient is of child bearing age,
* (f) patients with moderate or severe hepatic impairment
* (g) hemoglobin values less than 10% of the lower limit of normal per laboratory standards
* (h) inability to discontinue vasodilator treatment including calcium channel blockers, nitrates, alpha blockers, PDE-5 inhibitors, ACE inhibitors and angiotensin receptor blockers at least one week prior to the study,
* (i) echocardiographic evidence of pulmonary arterial hypertension [estimated right ventricular systolic pressure <35 mm Hg],
* (j) based on section 7.3 of the full prescribing information booklet- patients on cyclosporine, rifampin or ritonavir should be excluded,
* (k) patients with diffuse disease,
* (l) disease duration > 7 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NILANJANA BOSE, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Nilanjana Bose, Md, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Bose N, Bena J, Chatterjee S. Evaluation of the effect of ambrisentan on digital microvascular flow in patients with systemic sclerosis using laser Doppler perfusion imaging: a 12-week randomized double-blind placebo controlled trial. Arthritis Res Ther. 2015 Mar 5;17(1):44. doi: 10.1186/s13075-015-0558-9. PMID 25876611

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ambrisentan | Sugar Pill
Started | 15 | 5
Completed | 15 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan | Sugar Pill | Total
Number analyzed (Participants) | 15 | 5 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.8) | 46.8 (10.5) | 49.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Digital Micro-vascular Flow
Description: Change in digital micro-vascular flow measured by LDPI in patients with Raynaud's phenomenon (RP) and digital ischemia secondary to SSc at 1 week and 12 weeks
Time Frame: Baseline and 12 weeks
Population: Assuming a standard deviation of 0.40, and use of a two-sample t-test with significance level of 0.05, there will be 80% power to detect differences in the change from baseline of at least 0.65 units if moderate correlation (r=0.50) exists, and 0.45 units if strong correlation (r=0.75) exists between treated
Measure: Mean (95% Confidence Interval); unit: perfusion unit
Groups:
- Ambrisentan: Ambrisentan 5 mg daily for 1 month, then 10 mg daily for 2 months
- Sugar Pill: Placebo, same appearing as Ambrisentan
Arm/Group | Ambrisentan | Sugar Pill
Number analyzed (Participants) | 15 | 5
perfusion unit
  1 week | .11 [-0.15 to 0.37] | .18 [-.27 to .63]
  12 weeks | -.01 [-0.28 to .25] | -.06 [-0.51 to .39]

ADVERSE EVENTS:
Arm/Group | Ambrisentan | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5

LIMITATIONS AND CAVEATS:
Small sample size and short duration of study Some patients had hand contractures which made the LDPI images somewhat inaccurate Could not adjust for all variables in final analysis Placebo effect reflected in patient responses to questionnaires

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No